CLINICAL TRIAL: NCT06690801
Title: Dead Space and Inhaled Nitric Oxide in Pediatric Acute Respiratory Distress Syndrome
Acronym: DiNO
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Anoopindar Bhalla, Medical Staff/USC Faculty CWR, Children's Hospital Los Angeles
Other Study IDs: CHLA-24-00209; R01HL173488 (NIH)
Record Dates: First submitted 2024-11-08; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Pediatrics; Mechanical Ventilation; Inhaled Nitric Oxide
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with moderate to severe ARDS

SUMMARY:
The goal of this observational study is to determine whether a marker of dead space (the end-tidal to alveolar dead space fraction [AVDSf]) is more strongly associated with mortality risk than markers of oxygenation abnormality (oxygenation index) and to determine whether dead space (AVDSf) is an important marker of heterogeneity in the inhaled nitric oxide (iNO) treatment effect for children with acute respiratory distress syndrome (ARDS).

The study aims are:

1. To validate AVDSf for risk stratification of mortality in pediatric ARDS
2. To determine if there is heterogeneity in treatment effect for iNO defined by AVDSf
3. To detect the association between AVDSf and microvascular dysfunction trajectory and whether iNO therapy modifies this association

This is a prospective, multicenter observational study of 1260 mechanically ventilated children with moderate to severe ARDS. In a subgroup of 450 children with severe ARDS, longitudinal blood samples will be obtained to measure plasma protein markers.

ELIGIBILITY:
Inclusion Criteria:

* Age >37 weeks corrected gestational age to 21 years, including adults lacking the capacity to consent.
* Within 72 hours of the start of invasive mechanical ventilation and meet the criteria for pediatric ARDS (new infiltrate on chest imaging and a known ARDS risk factor within 7 days of the onset of hypoxemia) and either meet criteria for moderate or severe pediatric ARDS between 4-72 hours of IMV (OI ≥ 8 or OSI ≥ 7.5) OR have an OI ≥ 20 or an OSI ≥ 14 x 15 minutes between 0-4 hours of IMV.
* Subgroup of children eligible for longituduinal Blood Collection: Children with severe PARDS (OI ≥ 16 or an OSI ≥ 12 between 4-72 hours of IMV) or those with an OI ≥ 20 or an OSI ≥ 14 for 15 minutes between 0-4 hours of IMV will be eligible for collection of longitudinal plasma samples.

Exclusion Criteria:

* Non-conventional invasive mechanical ventilation (i.e. High Frequency Oscillatory Ventilation, Airway Pressure Release Ventilation) at the time of ICU admission
* ECMO or iNO (or other inhaled pulmonary vasodilator therapy) at the time of ICU admission
* Significant lower airways obstruction (examination of ventilator and capnography waveforms by site study or medical team)
* Air leak >20% (endotracheal tube, tracheostomy tube, or thoracostomy tube)
* Home Invasive Mechanical Ventilation
* Cyanotic Congenital Heart Disease
* Previous enrollment in the DiNO study
* Do not resuscitate order at the time of pediatric ARDS diagnosis.
* Blood gas not obtained prior to initiation of ECMO, iNO, or non-conventional ventilation.

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with moderate to severe ARDS
Sampling Method: Probability Sample
Enrollment: 1260 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants that experience all-cause mortality within 28 days from start of invasive mechanical ventilation | From the start of invasive mechanical ventilation to 28 days
  28 day all-cause mortality

SECONDARY OUTCOMES:
Number of participants that experience all-cause mortality within 90 days from start of invasive mechanical ventilation | From the start of invasive mechanical ventilation to 90 days
  90 day all-cause mortality
28-Day Ventilator-Free Days | From the start of invasive mechanical ventilation to 28 days
  The number of days within the first 28 days of invasive mechanical ventilation for ARDS that a patient is alive and free of mechanical ventilation.
The days on invasive mechanical ventilation for survivors of ARDS | From the start of invasive mechanical ventilation to the end of invasive mechanical ventilation (or 90 days after the start of invasive mechanical ventilation if the patient is still on invasive mechanical ventilation at 90 days)
  The number of days that a patient that survives is on invasive mechanical ventilation (up to 90 days)
The number of non-pulmonary organ failure free days within the first 14 days of invasive mechanical ventilation | From the start of invasive mechanical ventilation to 14 days
  Organ failure criteria will be determined with the Pediatric Organ Dysfunction Information Update Mandate. We will identify the number of days in the first 14 days of ARDS that a patient is alive and without any non-pulmonary organ failures.
The number of non-pulmonary organ failures 21 days after the start of invasive mechanical ventilation | 21 days after the start of invasive mechanical ventilation
  Organ failure criteria will be determined with the Pediatric Organ Dysfunction Information Update Mandate. The number of non-pulmonary organ failures on day 21 after the start of invasive mechanical ventilation will be identified. Patients that experience mortality prior to 21 days will be considered to have failure of all non-pulmonary organs.
The number of non-pulmonary organ failures 28 days after the start of invasive mechanical ventilation | 28 days after the start of invasive mechanical ventilation
  Organ failure criteria will be determined with the Pediatric Organ Dysfunction Information Update Mandate. The number of non-pulmonary organ failures on day 28 after the start of invasive mechanical ventilation will be identified. Patients that experience mortality prior to 28 days will be considered to have failure of all non-pulmonary organs.
The number of non-pulmonary organs that newly meet failure criteria or have an increase in the severity of organ failure within the first 14 days of invasive mechanical ventilation | From the start of invasive mechanical ventilation to 14 days
  Organ failure criteria will be determined with the Pediatric Organ Dysfunction Information Update Mandate. We will identify the number of organs during the first 14 days of invasive mechanical ventilation that either have worsening of the severity of failure or new failure after the first day of invasive mechanical ventilation.
The development of renal failure within the first 14 days of invasive mechanical ventilation | From the start of invasive mechanical ventilation to 14 days
  Renal organ failure criteria will be determined with the Pediatric Organ Dysfunction Information Update Mandate. We will identify whether during the first 14 days of invasive mechanical ventilation there is new renal failure after the first day of invasive mechanical ventilation.
Non-pulmonary organ failure phenotypes that develop within the first 14 days of invasive mechanical ventilation | From the start of invasive mechanical ventilation to 14 days
  Organ failure criteria will be determined with the Pediatric Organ Dysfunction Information Update Mandate. We will identify 14-day non-pulmonary organ failure free phenotypes using clustering analyses.
Cumulative non-pulmonary organ failure severity in the first 14 days of invasive mechanical ventilation | From the start of invasive mechanical ventilation to 14 days
  Organ failure scores will be quantified daily with the Pediatric Logistic Organ Dysfunction (PELOD-2) score. Children that die will be assigned the maximum value. The score will be summed over the first 14 days of invasive mechanical ventilation.
The change in functional status score from baseline to hospital discharge | From baseline to hospital discharge (or 90 days after the start of invasive mechanical ventilation)
  The baseline functional status score and the intensive care unit discharge functional status score will be compared and new morbidities will be identified. If the patient is still in the hospital after 90 days of the start of invasive mechanical ventilation the functional status score at 90 days will be used rather than the functional status score at hospital discharge.
The change in pediatric overall performance score from baseline to hospital discharge | From baseline to hospital discharge (or 90 days after the start of invasive mechanical ventilation)
  The baseline pediatric overall performance score and the hospital discharge pediatric overall performance score will be compared and new morbidities will be identified. If the patient is still in the hospital after 90 days of the start of invasive mechanical ventilation the pediatric overall performance score at 90 days will be used rather than the pediatric overall performance score at hospital discharge.
The change in pediatric cerebral performance score from baseline to hospital discharge | From baseline to hospital discharge (or 90 days after the start of invasive mechanical ventilation)
  The baseline pediatric cerebral performance score and the hospital discharge pediatric cerebral performance score will be compared and new morbidities will be identified. If the patient is still in the hospital after 90 days of the start of invasive mechanical ventilation the pediatric cerebral performance score at 90 days will be used rather than the pediatric cerebral performance score at hospital discharge.
All-cause mortality or the use of extracorporeal membrane oxygenation (ECMO) therapy within 28 days after the start of invasive mechanical ventilation | From the start of invasive mechanical ventilation to 28 days
  Patients who experience mortality or use of ECMO within 28 days of the start of invasive mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Anoopindar M Bhalla, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (10):
- United States (10):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Denver, Colorado
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan / CS Mott Children's Hospital, Ann Arbor, Michigan
  - University of Nebraska Medical Center / Children's Hospital and Medical Center, Omaha, Nebraska
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital Baylor College of Medicine, Houston, Texas
  - American Family Children's Hospital / University of Wisconsin-Madison, Madison, Wisconsin
  - Children's Hospital of Wisconsin / Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Deidentified public use dataset will be created.
Time Frame: available in 2029